CLINICAL TRIAL: NCT01869348
Title: IMPACT: Inactivity Monitoring and Physical Activity Controlled Trial
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-071
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2015-05

CONDITIONS: Obesity; Cardiovascular Disease; Cancer; Diabetes; Sarcopenia
Keywords: Physical activity; Activity monitor; Technology; Obesity; Aging muscle
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Neoplasms; Diabetes Mellitus; Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait list control (No Intervention): This group will receive no intervention until after data collection for the randomized trial is completed. Then, they will receive the monitor intervention.
- Monitor intervention (Experimental): This arm will receive the monitor intervention, including provision of a wristband activity monitor and mini-tablet as well as weekly counseling phone calls
  Interventions: Behavioral: Monitor intervention

INTERVENTIONS:
Behavioral: Monitor intervention — Investigators will lend each participant 1 Jawbone Up activity monitor and 1 mini tablet device. Participants will receive weekly brief phone calls with counseling related to self-efficacy and self-regulation. The monitors will be programmed to provide "idle alerts" that vibrate when participants have reached a cut point for a bout of sedentary behavior (e.g., 30 minutes). Participants will monitor their progress using an app on the tablet that provides graphical feedback on physical activity and sedentary behavior.
  Arms: Monitor intervention

SUMMARY:
As individuals age, their physical activity decreases and sedentary time increases. Even small changes in these two behaviors can greatly decrease risks for several major health problems, including cardiovascular disease, diabetes, and many cancers. Studies that use pedometers to encourage walking have successfully increased physical activity, but do not address sedentary behaviors such as television watching. The investigators propose to use a novel pedometer-like device (Jawbone Up) that encourages both increased physical activity and decreased sedentary time. First, the investigators will recruit 10 adults to participate in a brief intervention for six weeks. They will wear the wrist-based activity monitor and use a mini-tablet device to see feedback on their activity and sedentary time. They will also receive brief counseling weekly. The investigators will use this first study to investigate the basic feasibility of the intervention materials. Next, the investigators will recruit 20 adults and randomize them to receive the intervention for 12 weeks or to a waiting list. Here, the investigators will test the intervention with refinements made based on participant responses from the first small study. Our primary outcomes will be measures of feasibility and acceptability across all parts of the study. The investigators hypothesize that the intervention will be feasible and acceptable to the participants. The investigators will also measure physical activity, sedentary behavior, fitness, body fat, and psychological feelings of motivation.

DETAILED DESCRIPTION:
Inadequate physical activity and extended bouts of sedentary time are prevalent in adults, increasing from middle age into older adulthood. Even small changes in behavior, such as standing or walking in place periodically to break up sedentary bouts, can have large effects on cardiometabolic risk factors. Pedometer-based walking interventions have demonstrated effectiveness in increasing physical activity in this population, but these interventions have not targeted sedentary behavior. Recent technological advances have produced activity monitors that are capable of intervening on both behaviors. These wrist-worn monitors provide feedback and motivation for walking as well as cues to action in the form of idle alerts. These idle alerts vibrate when the wearer has remained sedentary for an extended period of time. Several preliminary studies have shown that older adults are willing to break up their sedentary time if prompted, but interventions thus far have relied upon television commercials as a cue to action. Use of these monitors would allow idle alerts to occur throughout the day, not only during television watching periods. The purpose of the IMPACT study (Inactivity Monitoring and Physical Activity Controlled Trial) is to investigate the feasibility of using activity monitors to simultaneously target both physical activity and sedentary behavior. First, we will conduct a pre-pilot test (N = 10) over six weeks. This brief study will provide basic feasibility and acceptability information on the monitor, content for weekly sessions, and assessments. Results will be used to refine the intervention for use in a larger pilot two-arm randomized controlled trial (N = 20, 12 weeks). This trial, comparing the intervention to a wait-list control group, will test feasibility, acceptability, and health, behavioral, and psychological outcomes. The primary outcome will be physical activity, operationalized as objectively-measured minutes of moderate-vigorous intensity physical activity over seven days (SenseWear armband). We will also measure cardiorespiratory fitness, physical function, body composition, and psychosocial variables such as autonomous motivation. The results of this innovative project will provide a foundation for future intervention in sedentary behavior and potentially create a large public health impact in a population at unique risk.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to be randomized to either group

Exclusion Criteria:

1. Age below 55 or above 79
2. Unable to read and understand English
3. Unable to read words in standard applications on a mobile device 5 - 10" large
4. Unable to find transportation to the study location
5. Investigator overseeing initial fitness test does not approve participation in the study
6. Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q, items 1 - 4). Reporting taking medicine for blood pressure on this questionnaire will require a doctor's note to participate.
7. Unable to walk for exercise (self-report)
8. Report current symptoms of alcohol or substance dependence
9. Plans to move away from the Galveston-Houston area or to be out of town for more than 1 week during the study period
10. Unwillingness to report drugs taken for comorbidities such as hypertension or diabetes
11. Stroke, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
12. Participant is active (60 minutes of moderate-vigorous intensity activity per week or more)
13. Participant watches little television (120 minutes per day or less)
14. BMI is under 25 kg/m2 or over 35 kg/m2
15. Another member of the household is a participant or staff member on this trial
16. Currently a participant in a physical activity research trial
17. Recently (less than six months ago) completed a physical activity research trial
18. Report a history of orthopedic complications that would prevent optimal participation in the physical activities prescribed (e.g., heel spurs, severe arthritis - may be eligible, but a doctor's note will be required)
19. Current smoker
20. Currently uses a Jawbone Up or similar activity monitor device

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Lyons, PhD, MPH, Principal Investigator — The University of Texas Medical Branch
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Lewis ZH, Swartz MC, Martinez E, Lyons EJ. Social Support Patterns of Middle-Aged and Older Adults Within a Physical Activity App: Secondary Mixed Method Analysis. JMIR Aging. 2019 Aug 23;2(2):e12496. doi: 10.2196/12496. PMID 31518281
- [Derived] Lyons EJ, Swartz MC, Lewis ZH, Martinez E, Jennings K. Feasibility and Acceptability of a Wearable Technology Physical Activity Intervention With Telephone Counseling for Mid-Aged and Older Adults: A Randomized Controlled Pilot Trial. JMIR Mhealth Uhealth. 2017 Mar 6;5(3):e28. doi: 10.2196/mhealth.6967. PMID 28264796

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wait List Control | Monitor Intervention
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait List Control | Monitor Intervention | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.70 (6.26) | 61.25 (5.00) | 61.48 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 13 | 13 | 26
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity From Baseline to 12 Weeks
Description: Minutes of physical activity measured over a seven day period
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wait List Control | Monitor Intervention
Number analyzed (Participants) | 20 | 20
minutes | -2.25 (33.91) | 50.93 (128.34)

2. Secondary Outcome: Change in Sedentary Behavior From Baseline to 12 Weeks
Description: Minutes of total sedentary time measured over a seven day period
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change in Autonomous Motivation From Baseline to 12 Weeks
Description: We will measure feelings of autonomous and controlled motivation/regulation for physical activity
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change in Physical Fitness From Baseline to 12 Weeks
Description: We will use the six minute walk test to measure physical fitness
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change in Body Composition From Baseline to 12 Weeks
Description: We will use dual x-ray absorptiometry (DEXA) to measure body composition, including body fat percentage and lean mass
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change in Physical Function From Baseline to 12 Weeks
Description: Functional measurements will be made using the Senior Fitness Test
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change in Weight From Baseline to 12 Weeks
Description: We will measure weight (and height at baseline) using a calibrated scale
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Feasibility
Description: We will use many different measures of feasibility, including adherence to study protocol, attrition, barriers to adherence, exposure/dose of intervention received, and any adverse events that occur
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Acceptability
Description: Acceptability will be self-reported using a variety of items taken from previous studies of physical activity interventions and usability
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Wait List Control | Monitor Intervention
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wait List Control (N=40) | Monitor Intervention (N=40)
Stitches to hand (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nerve damage during blood draw (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weakness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone spur (General disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes